CLINICAL TRIAL: NCT06533007
Title: The Role of Phosphodiesterase 3B in the Regulation of Human Adipose Tissue Biology and Systemic Glucose and Lipid Homeostasis
Brief Title: PDE3B in Metabolic Regulation
Status: Enrolling by invitation | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Maria Chondronikola, Principal Investigator and Lead for Human Nutrition, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: 343566
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Cardiometabolic Syndrome; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples and adipose tissue biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDE3B LoF group: Individuals heterozygous for a loss-of-function variant in the PDE3B gene
- Wild type group: Individuals who do not carry the loss-of-function variant for PDE3B gene but otherwise matched for age, sex, race/ethnicity, and body fat percent.

SUMMARY:
Phosphodiesterase 3B (PDE3B), an enzyme responsible for the degradation of cyclic AMP and GMP (two important second messengers used for intracellular signal transduction), has been associated with cardiometabolic outcomes. Results from animal studies indicate that abolishing PDE3B function may be associated with unfavourable metabolic profile; however, preliminary human studies suggest that heterozygous loss of function (LoF) variants in the PDE3B gene have been associated with cardiometabolic improvements. Therefore, the effect of PDE3B on human adipose tissue metabolic pathways remains poorly understood.

Accordingly, the investigators propose to conduct a recall-by-genotype, case-control study in a group of people with LoF variants in the PDE3B gene and a matched group without the variant (wild type, WT) to determine differences on key metabolic features: 1) adipose tissue biology (i.e., mitochondrial function, adipocyte morphology, gene expression and in vivo lipolysis in the basal and/or the insulin-stimulated state); 2) systemic lipid and glucose metabolism using the hyperinsulinemic-euglycemic clamp procedure.

The proposed investigations will elucidate the role of PDE3B on adipose tissue and systemic glucose and lipid metabolism in humans and whether modulating PDE3B activity constitutes a target for the prevention and treatment of cardiometabolic disease.

DETAILED DESCRIPTION:
Phosphodiesterase 3B (PDE3B) is a protein that plays a role in how cells handle nutrients (i.e. glucose and fats). The investigators have recently found that people who have a gene variant (i.e., change in the DNA) that reduces the function of the PDE3B protein may be protected from the development of diabetes and heart disease. However, it is unclear how this happens.

The aims of this study are to examine:

* What is the role of PDE3B in fat tissue function?
* How does PDE3B influence the way one's body handles blood sugars and lipids?

To this end, the investigators propose to study people who have a variant that reduces the function of that PDE3B and an equal number of people with the typical genotype.

Participants will be asked to attend two visits:

* a 4-h screening visit: involving a medical examination, blood tests before/after drinking a sugary drink and assessment of lifestyle (physical activity/sleep/diet) using questionnaires and smartwatch.
* a 24-h metabolic testing visit (only for eligible participants): involving an infusion of insulin and collection of blood samples and fat tissue from the lower tummy.

These investigations will provide a great opportunity to study how people with or without the variant handle fat, sugars and lipids in their bodies. They will also help the scientific community to understand the role of PDE3B in humans and possibly develop new ways to prevent or fight conditions like diabetes and heart disease.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to give informed consent for participation in the study
* aged 21-75 years
* men and women

Exclusion Criteria:

* unstable weight (>5% change the last 2 months)
* type 2 diabetes or other major organ dysfunction
* cancer in last 5 years
* gastrointestinal or bariatric surgery (except cholecystectomy and appendectomy)
* conditions that render subject unable to complete all testing procedures (including individuals with known allergies or contraindications to the medications used in this study)
* use of medications that affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued
* smoking
* illegal drug use
* pregnant or lactating
* unable to grant voluntary informed consent or comply with the study instructions

Ages: 21 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with heterozygous for PDE3B LoF variants will be recruited from existing research cohorts (i.e., the Oxford Biobank, the NIHR BioResource at the University of Cambridge and the Fenland study populations (1:700 frequency of the LoF variant). Subsequently, individuals without the variant of interest will be recruited from the same cohorts to establish a WT group of individuals matched for age, sex, race/ethnicity, and body fat percent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Lipolysis | baseline
  Lipolysis will be assessed as the palmitate rate of appearance by using infusion of stable isotope tracers.

SECONDARY OUTCOMES:
Adipose tissue gene expression | baseline
  Changes in the expression of genes will be assessed by using RNA sequencing
Insulin sensitivity | baseline
  Insulin sensitivity will be assessed by using a hyperinsulinemic euglycemic clamp procedure in conjunction with infusion of stable isotope tracers.
Insulin secretion | baseline
  Insulin sensitivity will be assessed by using an oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospital, Cambridge, United Kingdom